CLINICAL TRIAL: NCT01831427
Title: A Phase 1 Double-blind, Randomized, Placebo-Controlled, Staggered, Single and Multiple Ascending Dose, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of GS-5745 in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of GS-5745 (Andecaliximab) in Adults With Moderate to Severe Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-326-0101; 2013-000305-23 (EudraCT Number)
Record Dates: First submitted 2013-04-08; First posted 2013-04-15 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — andecaliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Andecaliximab 0.3 mg/kg IV single ascending dose (SAD) (Experimental): Participants will receive andecaliximab 0.3 milligrams per kilogram (mg/kg) on Day 1.
  Interventions: Drug: Andecaliximab
- Andecaliximab 1.0 mg/kg IV (SAD) (Experimental): Participants will receive andecaliximab 1.0 mg/kg on Day 1.
  Interventions: Drug: Andecaliximab
- Andecaliximab 2.5 mg/kg IV (SAD) (Experimental): Participants will receive andecaliximab 2.5 mg/kg on Day 1.
  Interventions: Drug: Andecaliximab
- Andecaliximab 5.0 mg/kg IV (SAD) (Experimental): Participants will receive andecaliximab 5.0 mg/kg on Day 1.
  Interventions: Drug: Andecaliximab
- Placebo Pooled (SAD) (Placebo Comparator): Participants will receive placebo on Day 1.
  Interventions: Drug: Placebo to match Andecaliximab
- Andecaliximab 0.3 mg/kg IV multiple ascending doses (MAD) (Experimental): Participants will receive andecaliximab 0.3 mg/kg on Days 1, 15, and 29.
  Interventions: Drug: Andecaliximab
- Andecaliximab 1.0 mg/kg IV (MAD) (Experimental): Participants will receive andecaliximab 1.0 mg/kg on Days 1, 15, and 29.
  Interventions: Drug: Andecaliximab
- Andecaliximab 2.5 mg/kg IV (MAD) (Experimental): Participants will receive andecaliximab 2.5 mg/kg on Days 1, 15, and 29.
  Interventions: Drug: Andecaliximab
- Andecaliximab 5.0 mg/kg IV (MAD) (Experimental): Participants will receive andecaliximab 5.0 mg/kg on Days 1, 15, and 29.
  Interventions: Drug: Andecaliximab
- Andecaliximab 150 mg SC (Adaptive MAD) (Experimental): Participants will receive andecaliximab 150 mg on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: Andecaliximab
- Placebo Pooled (MAD) (Placebo Comparator): Participants will receive placebo on Days 1, 15, and 29.
  Interventions: Drug: Placebo to match Andecaliximab

INTERVENTIONS:
Drug: Andecaliximab — Andecaliximab administered by intravenous (IV) infusion or subcutaneous (SC) injection
  Other Names: GS-5745
  Arms: Andecaliximab 0.3 mg/kg IV multiple ascending doses (MAD); Andecaliximab 0.3 mg/kg IV single ascending dose (SAD); Andecaliximab 1.0 mg/kg IV (MAD); Andecaliximab 1.0 mg/kg IV (SAD); Andecaliximab 150 mg SC (Adaptive MAD); Andecaliximab 2.5 mg/kg IV (MAD); Andecaliximab 2.5 mg/kg IV (SAD); Andecaliximab 5.0 mg/kg IV (MAD); Andecaliximab 5.0 mg/kg IV (SAD)
Drug: Placebo to match Andecaliximab — Placebo to match andecaliximab administered by IV infusion
  Arms: Placebo Pooled (MAD); Placebo Pooled (SAD)

SUMMARY:
The primary objectives of this study are as follows:

* To assess the safety and tolerability of escalating single and multiple doses of GS-5745 (andecaliximab) in participants with moderate to severe ulcerative colitis (UC) as assessed by adverse events (AEs) and laboratory abnormalities
* To assess the pharmacokinetics (PK) of GS-5745 (andecaliximab) in participants with moderate to severe UC.

DETAILED DESCRIPTION:
The study will test the safety of the drug. Participants will be given different concentrations of the drug in Cohorts, starting from a lower dose to a higher dose.

Single-Dose Treatment:

A thorough assessment of safety and tolerability will be performed before escalating to the next higher dose. For example, the first 2 participants will be dosed in a staggered fashion 24 hours apart. Provided that there are no significant safety signals up to 24 hours post-dose for the first 2 participants, the remaining 4 participants will be dosed. A thorough assessment of safety and tolerability (through Day 14 post-dose) will be performed by the safety review committee before escalating to the next higher dose. Participants enrolled in a SAD cohort will be eligible to participate in a MAD or adaptive MAD cohort if eligibility criteria are met.

Multiple-Dose Treatment:

This design follows the same set-up as the Single-Dose Treatment. Dosing will not commence in the first MAD cohort until safety data from the second dose level SAD cohort has been reviewed through Day 15. Successive MAD cohorts will only be dosed after safety data from the previous, lower dose MAD cohort through Day 43 and the next higher dose SAD cohort through Day 15, have been reviewed by the safety review committee. An additional Adaptive MAD cohort will explore a subcutaneous dosing of andecaliximab 150 mg prefilled syringe once a week for 5 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or Female, 18 to 65 years of age
* Negative pregnancy test at screening
* Documented diagnosis of UC with a minimum disease extent of 15 centimeters (cm) from the anal verge
* Mayo Score of at least 3 for the SAD cohort and Mayo Score of at least 6 for the MAD cohorts
* Hepatic panel (aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, direct bilirubin, alkaline phosphatase, lactate dehydrogenase [LDH] ≤ 2 times the upper limit of the normal range [ULN])
* Serum creatinine ≤ 1.5 times the ULN
* Hemoglobin ≥ 10 grams per deciliter (g/dL) (both males and females)
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1,500 milli meters [mm]^3)
* Platelets ≥ 100 x 10^9/L.

Key Exclusion Criteria:

* Pregnant or lactating females
* Exhibit severe UC/ clinically significant active infection
* Current use of oral corticosteroids at a dose equivalent to > 20 mg/day of prednisone
* Any dose adjustment in oral corticosteroids or oral immunosuppressants (6-MP, Azathioprine), or oral 5-aminosalicylate (5-ASA) compounds within 30 days of Baseline
* Use of rectal formulations of 5-ASA compounds or corticosteroids within 2 weeks prior to randomization
* Crohn's disease or indeterminate colitis
* History of colectomy, partial colectomy, or dysplasia on biopsy
* Stool sample positive for Clostridium difficile (C. difficile) toxin, E. coli, Salmonella, Shigella, Campylobacter or Yersinia
* Treatment with Infliximab, Adalimumab, Natalizumab, Golimumab, Vedolizumab or Certolizumab within 8 weeks of randomization
* Any chronic medical condition (including, but not limited to, cardiac or pulmonary disease) that, in the opinion of the Investigator, would make the individual unsuitable for the study or would prevent compliance with the study protocol.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2015-01-05 (Actual); Study Completion 2015-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- United States (6):
  - Delta Research Partners LLC, Monroe, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Clinical Research Institute of Michigan, Chesterfield Township, MI 48047, Michigan
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Community Research, Cincinnati, Ohio
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - GIRI, Vancouver, British Columbia
  - LHSC University Campus, London, Ontario
- Hungary (3):
  - Clinical Pharma Center of Kenezy Gyula Korhaz Rendelointezet, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest, Pest County
  - Drug Research Centre, Balatonfüred
- Republican Clinical Hospital, Chisinau, Moldova
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
- Institute of Pulmonology "Marius Nasta", Bucharest, Romania

REFERENCES:
- [Result] Bhandari BR, Fogel R, Onken J, Yen EH, Kanwar B, Subramanian GM, McHutchison GJ, et al. Safety and Efficacy of GS-5745 an Anti-Matrix Metalloproteinase 9 (MMP) Monoclonal Antibody in Patients with Moderately to Severely Active Ulcerative Colitis. Gastroenterology 2015;148 (4): S-1196.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, and Europe. The first participant was screened on 28 March 2013. The last study visit occurred on 06 February 2015.
Pre-assignment Details: 124 participants were screened.
Groups:
- Andecaliximab 0.3 mg/kg IV Single Ascending Dose (SAD): Participants received a single intravenous (IV) infusion of andecaliximab 0.3 milligrams per kilogram (mg/kg) on Day 1.
- Andecaliximab 1.0 mg/kg IV (SAD): Participants received a single IV infusion of andecaliximab 1.0 mg/kg on Day 1.
- Andecaliximab 2.5 mg/kg IV (SAD): Participants received a single IV infusion of andecaliximab 2.5 mg/kg on Day 1.
- Andecaliximab 5.0 mg/kg IV (SAD): Participants received a single IV infusion of andecaliximab 5.0 mg/kg on Day 1.
- Placebo Pooled (SAD): Participants received a single IV infusion of placebo on Day 1.
- Andecaliximab 0.3 mg/kg IV Multiple Ascending Doses (MAD): Participants received 3 single IV infusions of andecaliximab 0.3 mg/kg on Days 1, 15, and 29.
- Andecaliximab 1.0 mg/kg IV (MAD): Participants received 3 single IV infusions of andecaliximab 1.0 mg/kg on Days 1, 15, and 29.
- Andecaliximab 2.5 mg/kg IV (MAD): Participants received 3 single IV infusions of andecaliximab 2.5 mg/kg on Days 1, 15, and 29.
- Andecaliximab 5.0 mg/kg IV (MAD): Participants received 3 single IV infusions of andecaliximab 5.0 mg/kg on Days 1, 15, and 29.
- Andecaliximab 150 mg SC (Adaptive MAD): Participants received 5 single subcutaneous (SC) doses of andecaliximab 150 mg on Days 1, 8, 15, 22, and 29.
- Placebo Pooled (MAD): Participants received 3 single IV infusions of placebo on Days 1, 15, and 29.
Period: Overall Study
Arm/Group | Andecaliximab 0.3 mg/kg IV Single Ascending Dose (SAD) | Andecaliximab 1.0 mg/kg IV (SAD) | Andecaliximab 2.5 mg/kg IV (SAD) | Andecaliximab 5.0 mg/kg IV (SAD) | Placebo Pooled (SAD) | Andecaliximab 0.3 mg/kg IV Multiple Ascending Doses (MAD) | Andecaliximab 1.0 mg/kg IV (MAD) | Andecaliximab 2.5 mg/kg IV (MAD) | Andecaliximab 5.0 mg/kg IV (MAD) | Andecaliximab 150 mg SC (Adaptive MAD) | Placebo Pooled (MAD)
Started | 5 | 5 | 5 | 5 | 4 | 8 | 8 | 8 | 8 | 10 | 8
Completed | 5 | 4 | 5 | 4 | 4 | 7 | 6 | 7 | 8 | 9 | 5
Not Completed | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Not completed — Investigator's Discretion | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Groups:
- Andecaliximab 0.3 mg/kg IV (SAD): Participants received a single IV infusion of andecaliximab 0.3 mg/kg on Day 1.
- Andecaliximab 0.3 mg/kg IV (MAD): Participants received 3 single IV infusions of andecaliximab 0.3 mg/kg on Days 1, 15, and 29.
- Andecaliximab 150 mg SC (Adaptive MAD): Participants received 5 single SC doses of andecaliximab 150 mg on Days 1, 8, 15, 22, and 29.
- Total: Total of all reporting groups
Arm/Group | Andecaliximab 0.3 mg/kg IV (SAD) | Andecaliximab 1.0 mg/kg IV (SAD) | Andecaliximab 2.5 mg/kg IV (SAD) | Andecaliximab 5.0 mg/kg IV (SAD) | Placebo Pooled (SAD) | Andecaliximab 0.3 mg/kg IV (MAD) | Andecaliximab 1.0 mg/kg IV (MAD) | Andecaliximab 2.5 mg/kg IV (MAD) | Andecaliximab 5.0 mg/kg IV (MAD) | Andecaliximab 150 mg SC (Adaptive MAD) | Placebo Pooled (MAD) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 8 | 8 | 8 | 8 | 10 | 8 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11.3) | 37 (11.3) | 45 (15.4) | 42 (12.9) | 41 (15.1) | 42 (13.9) | 39 (11.7) | 38 (13.7) | 50 (9.8) | 48 (8.8) | 44 (15.8) | 43 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 3 | 3 | 5 | 3 | 5 | 2 | 6 | 3 | 38
  Male | 1 | 2 | 4 | 2 | 1 | 3 | 5 | 3 | 6 | 4 | 5 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 5 | 4 | 8 | 8 | 8 | 8 | 10 | 8 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not permitted means not permitted to ask due to local regulations.
  Participants
    Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race: Asian | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Race: Black | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 8
    Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race: White | 2 | 3 | 5 | 5 | 3 | 7 | 7 | 8 | 8 | 8 | 8 | 64
    Race: Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race: Not Permitted | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Any Treatment-Emergent Adverse Events (TEAEs) (SAD/MAD)
Description: TEAEs are any AEs with an onset date of on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug or any AEs leading to premature discontinuation of study drug.
Time Frame: SAD Cohorts: First dose date (Day 1) plus 30 days, MAD/Adaptive MAD Cohort: First dose date up to last dose date (Maximum: Day 29) plus 30 days
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Andecaliximab IV Combined (SAD): Participants who received a single IV infusion of andecaliximab (0.3, 1.0, 2.5 and 5.0 mg/kg on Day 1) were combined in this arm.
- Andecaliximab IV Combined (MAD): Participants who received 3 single IV infusions of andecaliximab (0.3, 1.0, 2.5, 5.0 mg/kg on Days 1, 15, and 29) were combined in this arm.
- Andecaliximab IV+SC Combined (MAD): Participants who received 3 single IV infusions of andecaliximab (0.3, 1.0, 2.5, 5.0 mg/kg on Days 1, 15, and 29) and 5 single SC dose of andecaliximab (150 mg on Days 1, 8, 15, 22, and 29) were combined in this arm.
Arm/Group | Andecaliximab 0.3 mg/kg IV (SAD) | Andecaliximab 1.0 mg/kg IV (SAD) | Andecaliximab 2.5 mg/kg IV (SAD) | Andecaliximab 5.0 mg/kg IV (SAD) | Andecaliximab IV Combined (SAD) | Placebo Pooled (SAD) | Andecaliximab 0.3 mg/kg IV (MAD) | Andecaliximab 1.0 mg/kg IV (MAD) | Andecaliximab 2.5 mg/kg IV (MAD) | Andecaliximab 5.0 mg/kg IV (MAD) | Andecaliximab IV Combined (MAD) | Andecaliximab 150 mg SC (Adaptive MAD) | Andecaliximab IV+SC Combined (MAD) | Placebo Pooled (MAD)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20 | 4 | 8 | 8 | 8 | 8 | 32 | 10 | 42 | 8
percentage of participants | 0.0 | 20.0 | 20.0 | 60.0 | 25.0 | 25.0 | 25.0 | 75.0 | 62.5 | 62.5 | 56.3 | 50.0 | 54.8 | 62.5

2. Primary Outcome: Pharmacokinetic (PK) Parameter: Cmax (SAD)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Predose and 1, 2, and 6 hours postdose on Day 1; Days 2, 3, 8, 15, 29, and 43
Population: Participants in the PK Analysis Set (who received at least 1 dose of study drug and had at least 1 non-missing post dose concentration value for the corresponding analyte in plasma) for the SAD cohorts were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Andecaliximab 0.3 mg/kg IV (SAD) | Andecaliximab 1.0 mg/kg IV (SAD) | Andecaliximab 2.5 mg/kg IV (SAD) | Andecaliximab 5.0 mg/kg IV (SAD)
Number analyzed (Participants) | 5 | 5 | 5 | 5
micrograms per milliliter (μg/mL) | 9.4 (3.28) | 32.7 (11.08) | 77.8 (20.67) | 210.0 (102.60)

3. Primary Outcome: PK Parameter: Cmax (MAD)
Description: Cmax is defined as the maximum concentration of drug over the dosing interval. Data for Day 1 was based on the data collected from Day 1 through Day 8. Data for Day 29 was based on the data collected from Day 29 through Day 36.
Time Frame: MAD Cohorts: Predose and 1, 2, and 6 hours postdose on Days 1 and 29, Predose on Days 8 and 36; Adaptive MAD Cohort: Predose and 6 hours postdose on Days 1, and 29, Predose on Days 8 and 36
Population: Participants in the PK Analysis Set for MAD cohort (with available data) and Adaptive MAD cohort were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Andecaliximab 0.3 mg/kg IV (MAD) | Andecaliximab 1.0 mg/kg IV (MAD) | Andecaliximab 2.5 mg/kg IV (MAD) | Andecaliximab 5.0 mg/kg IV (MAD) | Andecaliximab 150 mg SC (Adaptive MAD)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9
μg/mL
  Day 1 | 9.0 (3.23) | 33.7 (26.43) | 57.1 (13.66) | 95.3 (28.93) | NA (NA) — Not evaluated at Day 1 for the andecaliximab 150 mg SC group.
  Day 29: number analyzed (Participants) | 7 | 8 | 8 | 8 | 9
  Day 29 | 10.3 (5.06) | 29.0 (10.89) | 66.6 (15.02) | 120.8 (21.15) | 33.5 (42.47)

4. Primary Outcome: PK Parameter: Ctau (MAD)
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: MAD Cohorts: Predose and 1, 2, and 6 hours postdose on Day 29; Predose on Day 36; Adaptive MAD Cohort: Predose and 6 hours postdose on Day 29; Predose on Day 36
Population: Participants in the PK Analysis Set for MAD and Adaptive MAD cohorts were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Andecaliximab 0.3 mg/kg IV (MAD) | Andecaliximab 1.0 mg/kg IV (MAD) | Andecaliximab 2.5 mg/kg IV (MAD) | Andecaliximab 5.0 mg/kg IV (MAD) | Andecaliximab 150 mg SC (Adaptive MAD)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 9
μg/mL | NA (NA) — Values were all below the limit of quantitation. | NA (NA) — Values were all below the limit of quantitation. | 0.8 (2.36) | 27.2 (13.99) | 16.0 (15.99)

5. Primary Outcome: PK Parameter: AUCinf (SAD)
Description: AUCinf is defined as the area under the plasma concentration versus time curve extrapolated to infinite time.
Time Frame: Predose and 1, 2, and 6 hours postdose on Day 1; Days 2, 3, 8, 15, 29, and 43
Population: Participants in the PK Analysis Set for SAD cohorts were analyzed.
Measure: Mean (Standard Deviation); unit: day*micrograms per milliliter(day*μg/mL)
Arm/Group | Andecaliximab 0.3 mg/kg IV (SAD) | Andecaliximab 1.0 mg/kg IV (SAD) | Andecaliximab 2.5 mg/kg IV (SAD) | Andecaliximab 5.0 mg/kg IV (SAD)
Number analyzed (Participants) | 5 | 5 | 5 | 5
day*micrograms per milliliter(day*μg/mL) | 9.4 (4.44) | 66.6 (22.85) | 240.8 (23.69) | 817.3 (405.97)

6. Primary Outcome: PK Parameter: AUCtau (MAD)
Description: AUCtau is defined as the area under the plasma concentration versus time curve over the dosing interval. Data for Day 1 was based on the data collected from Day 1 through Day 8. Data for Day 29 was based on the data collected from Day 29 through Day 36.
Time Frame: MAD Cohorts: Predose and 1, 2, and 6 hours postdose on Days 1 and 29; Predose on Days 8 and 36; Adaptive MAD Cohort: Predose and 6 hours postdose on Days 1, and 29; Predose on Days 8 and 36
Population: Participants in the PK Analysis Set for MAD and Adaptive MAD cohorts with available data were analyzed. Concentrations fell below the limit of quantitation early in the dosing interval for some participants in some of the cohorts. Therefore, AUCtau couldn't be adequately estimated and was not included.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Andecaliximab 0.3 mg/kg IV (MAD) | Andecaliximab 1.0 mg/kg IV (MAD) | Andecaliximab 2.5 mg/kg IV (MAD) | Andecaliximab 5.0 mg/kg IV (MAD) | Andecaliximab 150 mg SC (Adaptive MAD)
Number analyzed (Participants) | 7 | 5 | 6 | 8 | 9
day*μg/mL | NA (NA) — Concentrations in this group fell below the limit of quantitation early in the dosing interval. Therefore, AUCtau couldn't be adequately estimated for all participants. | 79.2 (53.98) | 251.8 (88.15) | 784.8 (262.5) | 166.8 (164.53)

7. Primary Outcome: PK Parameter: AUClast (SAD)
Description: AUClast is defined as the area under the plasma concentration versus time curve from time zero to the last observable concentration.
Time Frame: Predose and 1, 2, and 6 hours postdose on Day 1; Days 2, 3, 8, 15, 29, and 43
Population: Participants in the PK Analysis Set for SAD cohorts were analyzed.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Andecaliximab 0.3 mg/kg IV (SAD) | Andecaliximab 1.0 mg/kg IV (SAD) | Andecaliximab 2.5 mg/kg IV (SAD) | Andecaliximab 5.0 mg/kg IV (SAD)
Number analyzed (Participants) | 5 | 5 | 5 | 5
day*μg/mL | 7.7 (2.54) | 57.2 (26.96) | 212.4 (38.79) | 750.2 (412.42)

ADVERSE EVENTS:
Time Frame: SAD Cohorts: First dose date (Day 1) plus 30 days, MAD/Adaptive MAD Cohort: First dose date up to last dose date (Maximum: Day 29) plus 30 days.
Description: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Arm/Group | Andecaliximab 0.3 mg/kg IV (SAD) | Andecaliximab 1.0 mg/kg IV (SAD) | Andecaliximab 2.5 mg/kg IV (SAD) | Andecaliximab 5.0 mg/kg IV (SAD) | Andecaliximab IV Combined (SAD) | Placebo Pooled (SAD) | Andecaliximab 0.3 mg/kg IV (MAD) | Andecaliximab 1.0 mg/kg IV (MAD) | Andecaliximab 2.5 mg/kg IV (MAD) | Andecaliximab 5.0 mg/kg IV (MAD) | Andecaliximab IV Combined (MAD) | Andecaliximab 150 mg SC (Adaptive MAD) | Andecaliximab IV+SC Combined (MAD) | Placebo Pooled (MAD)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/20 | 0/4 | 0/8 | 0/8 | 0/8 | 0/8 | 0/32 | 0/10 | 0/42 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 0/5 | 0/5 | 1/20 | 0/4 | 1/8 | 1/8 | 0/8 | 0/8 | 2/32 | 0/10 | 2/42 | 1/8
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 3/5 | 4/20 | 1/4 | 2/8 | 6/8 | 5/8 | 5/8 | 18/32 | 5/10 | 23/42 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab 0.3 mg/kg IV (SAD) (N=5) | Andecaliximab 1.0 mg/kg IV (SAD) (N=5) | Andecaliximab 2.5 mg/kg IV (SAD) (N=5) | Andecaliximab 5.0 mg/kg IV (SAD) (N=5) | Andecaliximab IV Combined (SAD) (N=20) | Placebo Pooled (SAD) (N=4) | Andecaliximab 0.3 mg/kg IV (MAD) (N=8) | Andecaliximab 1.0 mg/kg IV (MAD) (N=8) | Andecaliximab 2.5 mg/kg IV (MAD) (N=8) | Andecaliximab 5.0 mg/kg IV (MAD) (N=8) | Andecaliximab IV Combined (MAD) (N=32) | Andecaliximab 150 mg SC (Adaptive MAD) (N=10) | Andecaliximab IV+SC Combined (MAD) (N=42) | Placebo Pooled (MAD) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab 0.3 mg/kg IV (SAD) (N=5) | Andecaliximab 1.0 mg/kg IV (SAD) (N=5) | Andecaliximab 2.5 mg/kg IV (SAD) (N=5) | Andecaliximab 5.0 mg/kg IV (SAD) (N=5) | Andecaliximab IV Combined (SAD) (N=20) | Placebo Pooled (SAD) (N=4) | Andecaliximab 0.3 mg/kg IV (MAD) (N=8) | Andecaliximab 1.0 mg/kg IV (MAD) (N=8) | Andecaliximab 2.5 mg/kg IV (MAD) (N=8) | Andecaliximab 5.0 mg/kg IV (MAD) (N=8) | Andecaliximab IV Combined (MAD) (N=32) | Andecaliximab 150 mg SC (Adaptive MAD) (N=10) | Andecaliximab IV+SC Combined (MAD) (N=42) | Placebo Pooled (MAD) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 5 | 0 | 5 | 3
Wandering pacemaker (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 3 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 0 | 3 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.